CLINICAL TRIAL: NCT06437782
Title: Exploration of Health Literacy in Diabetes in Reunion Island and Metropolitan France
Brief Title: Exploration of Health Literacy in Diabetes in Reunion Island and France
Acronym: HLQ-Diabete
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de la Réunion (Other)
Responsible Party: Sponsor
Other Study IDs: 2017/CHU/13
Record Dates: First submitted 2024-05-22; First posted 2024-05-31 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Diabetes type1; Diabetes Type 2; Diabetes, Gestational
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes, Gestational

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- type 1 diabetes closed loop
  Interventions: Other: Questionnaire completion
- type 2 diabetes
  Interventions: Other: Questionnaire completion
- Gestational diabetes
  Interventions: Other: Questionnaire completion

INTERVENTIONS:
Other: Questionnaire completion — HLQ (Health Literacy questionnaire) will be completed by all included patients once.

SUMMARY:
The goal of this observational study is to identify the health literacy profile of diabetic patients in Reunion Island and France in order to obtain information to improve access to information, therapeutic education and to health service. The main question[s] it aims to answer [is/are]:

Participants will complete the Health Literacy Questionnaire (HLQ) once.

ELIGIBILITY:
Inclusion Criteria:

Patient with type 1, 2 or gestational diabetes taken care in hospital

Exclusion Criteria:

* Patient unable to understand and respect study procedures
* Patient with cognitive disorder
* Patient with serious acute complication due to diabetes within 15 days before inclusion
* Stroke history with neurologic consequences
* Other specific types of diabetes : chronic calcific pancreatitis, iatrogenic, other secondary diabetes, rare monogenic or genetic diabetes due to insulin resistance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with type 1 diabetes (strict insulin dependence, or anti-GAD, anti-IA2, and/or anti-ZnT8 + antibodies) with a hybrid closed-loop insulin therapy system for at least 3 months , diabetes of type 2 (non-insulin-dependent or insulin-requiring, with negative anti-GAD, anti-IA2, and/or anti-ZnT8 Ab if diabetes has been diagnosed for less than 5 years at the time of insulin therapy), or diabetes during pregnancy: gestational diabetes (diabetes diagnosed during pregnancy according to the diagnostic criteria of French recommendations), or pre-existing diabetes (known or not) with pregnancy.
Sampling Method: Non-Probability Sample
Enrollment: 1350 (Estimated)
Dates: Start 2025-04-17 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Health literacy profiles in Reunion Island | at inclusion
  HLQ (Health literacy questionnaire) is completed once. The algorithm produces unweighted scores for each of the 9 scales of the HLQ. The final score for each scale is an average score across all the questions that form that scale. The HLQ does not provide one overall summative score; rather it gives you nine separate scores that indicate a person's strengths and needs in relation to their health literacy.

SECONDARY OUTCOMES:
Health literacy profiles in Reunion Island and France | at inclusion
  HLQ (Health literacy questionnaire) is completed once. Health literacy profile in patients treated on Reunion Island et France will be described.
  The algorithm produces unweighted scores for each of the 9 scales of the HLQ. The final score for each scale is an average score across all the questions that form that scale. The HLQ does not provide one overall summative score; rather it gives you nine separate scores that indicate a person's strengths and needs in relation to their health literacy.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de La Réunion, Saint-Denis, Reunion

IPD SHARING:
Plan to Share IPD: No